CLINICAL TRIAL: NCT02796950
Title: The Effect of Acipimox on GLP-1 Secretion in Healthy Subjects: a Pilot Study
Brief Title: The Effect of Acipimox on GLP (Glucagon-like Peptide)-1 Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLP-1-16-02-261-16
Record Dates: First submitted 2016-05-27; First posted 2016-06-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Acipimox; GLP-1; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — acipimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acipimox (Experimental): Administration of acipimox 250 mg p.o.
  Interventions: Drug: Acipimox
- Control (No Intervention): No intervention.

INTERVENTIONS:
Drug: Acipimox — P.o. administration of 250 mg acipimox
  Other Names: Olbetam
  Arms: Acipimox

SUMMARY:
Glucagon like peptide 1 is produced in enteroendocrine L cells in the small intestine stimulated by peroral food intake. GLP-1 induces insulin secretion, and analogues are used in the treatment of DM2 (type 2 diabetes mellitus). Recently it was found, that levels of GLP-1 are increased in response to acipimox. The hypothesis is that G protein coupled receptors on enteroendocrine L cells bind acipimox and thereby induce GLP-1 secretion.

In a controlled, open, randomized experiment, eight healthy, overweight men will be studied on an intervention day, where they receive acipimox, and on a control day. The study day includes an OGTT (oral glucose tolerance test), blood samples before and after the OGTT and a biopsy from adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Adult men
* Healthy
* BMI 25-35

Exclusion Criteria:

* Known DM2
* Receiving hypolipidemic drugs

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Levels of GLP-1 in plasma | 9 months

SECONDARY OUTCOMES:
Lipolytic activity in adipose tissue by measuring FFA (free fatty acid) levels | 9 months
Insulin sensitivity by measuring blood glucose after an OGTT | 5 months

OTHER OUTCOMES:
Insulin secretion by measuring levels of insulin and c-peptid | 9 months
Secretion of the hormones ghrelin, leptin and GIP (gastric inhibitory polypeptide) by measuring hormone levels in plasma | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator — University of Aarhus
Locations (1):
- University Hospital of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pais R, Gribble FM, Reimann F. Stimulation of incretin secreting cells. Ther Adv Endocrinol Metab. 2016 Feb;7(1):24-42. doi: 10.1177/2042018815618177. PMID 26885360
- [Background] Iepsen EW, Torekov SS, Holst JJ. Liraglutide for Type 2 diabetes and obesity: a 2015 update. Expert Rev Cardiovasc Ther. 2015;13(7):753-67. doi: 10.1586/14779072.2015.1054810. PMID 26106933
- [Background] Tunaru S, Kero J, Schaub A, Wufka C, Blaukat A, Pfeffer K, Offermanns S. PUMA-G and HM74 are receptors for nicotinic acid and mediate its anti-lipolytic effect. Nat Med. 2003 Mar;9(3):352-5. doi: 10.1038/nm824. Epub 2003 Feb 3. PMID 12563315
- [Background] Newman JC, Verdin E. Ketone bodies as signaling metabolites. Trends Endocrinol Metab. 2014 Jan;25(1):42-52. doi: 10.1016/j.tem.2013.09.002. Epub 2013 Oct 18. PMID 24140022
- [Background] Fulcher GR, Walker M, Catalano C, Farrer M, Alberti KG. Acute metabolic and hormonal responses to the inhibition of lipolysis in non-obese patients with non-insulin-dependent (type 2) diabetes mellitus: effects of acipimox. Clin Sci (Lond). 1992 May;82(5):565-71. doi: 10.1042/cs0820565. PMID 1317767